CLINICAL TRIAL: NCT02917278
Title: Pilot Study of Nutrition in Maintenance Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Kathleen Hill Gallant, Assistant professor nutrition science, Purdue University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1510016673
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: End-Stage Renal Disease; Meals; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meals (Experimental): High-protein renal-specific meals
  Interventions: Dietary Supplement: Meals
- Control (No Intervention): No Meals

INTERVENTIONS:
Dietary Supplement: Meals — High Protein renal-specific meals
  Arms: Meals

SUMMARY:
This pilot study aims to produce preliminary data on the safety of providing high-protein meals to patients during dialysis, and effects of this intervention on nutritional status and quality of life outcomes. This is a non-randomized, parallel arm study. Meals provided will follow recommended dietary guidelines for HD patients and will provide approximately 1/3 of daily recommended protein intake. Patients will be allocated to either the treatment or control group by HD shift schedule. 2 months of baseline data will be collected, followed by 9 weeks of meal intervention/control and data collection. The primary outcome will be frequency of hypotensive events during dialysis requiring intervention. Secondary outcomes will include highest and lowest systolic blood pressure during dialysis, blood biochemistries including measures of renal function, nutritional status, and electrolyte balance; dialysis compliance; fluid retention; sleep and other quality of life measures; and dietary intake data.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Any race
* Age 18 years or older
* Maintenance hemodialysis patients

Exclusion Criteria:

• Patients with dysphagia that cannot be accommodated by texture modifications, or those exclusively NPO/requiring tube feeding or parenteral feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Hill Gallant, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participate data is available to other researchers upon reasonable request.

REFERENCES:
- [Result] Choi MS, Kistler B, Wiese GN, Stremke ER, Wright AJ, Moorthi RN, Moe SM, Hill Gallant KM. Pilot Study of the Effects of High-Protein Meals During Hemodialysis on Intradialytic Hypotension in Patients Undergoing Maintenance Hemodialysis. J Ren Nutr. 2019 Mar;29(2):102-111. doi: 10.1053/j.jrn.2018.06.002. Epub 2018 Aug 11. PMID 30107974
- Available data/document: Meeting abstract — https://www.asn-online.org/api/download/?file=/education/kidneyweek/archives/KW16Abstracts.pdf — Abstract presented as a poster at the ASN Kidney Week 2016 (TH-PO762)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Meals | Control
Started | 10 | 9
Completed | 9 | 9
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meals | Control | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (11.4) | 58.1 (19.2) | 62.4 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
Body Mass Index, kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 34.2 (10.2) | 31.1 (8.0) | 32.6 (9.0)
Years on Dialysis [Mean (Standard Deviation); unit: years] | 3.1 (2.0) | 3.6 (3.3) | 3.3 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Hypotensive Event Frequency
Description: frequency of hypotensive events that require intervention during dialysis
Time Frame: 9 weeks
Measure: Number; unit: events
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
events | 18 | 13

2. Secondary Outcome: Mean Arterial Pressure (mm Hg)
Description: Average Lowest Mean Arterial Pressure (mm Hg) over 25 dialysis sessions during the study.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
mm Hg | 75 (8) | 84 (11)

3. Secondary Outcome: Serum Albumin
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
g/dL | 3.7 (0.3) | 3.8 (0.3)

4. Secondary Outcome: Blood Urea Nitrogen
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
mg/dL | 49 (16) | 59 (13)

5. Secondary Outcome: Serum Creatinine
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
mg/dL | 6.8 (1.1) | 7.8 (4.4)

6. Secondary Outcome: Blood Glucose
Time Frame: 9 weeks
Population: Only measured in patients with diabetes mellitus
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Meals | Control
Number analyzed (Participants) | 8 | 6
mg/dL | 137 (55) | 178 (77)

7. Secondary Outcome: Serum Adjusted Calcium
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
mg/dL | 9.3 (0.4) | 9.3 (0.6)

8. Secondary Outcome: Serum Sodium
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
mEq/L | 138 (2) | 137 (3)

9. Secondary Outcome: Serum Phosphate
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
mg/dL | 5.2 (0.7) | 7.0 (1.7)

10. Secondary Outcome: Serum Chloride
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
mEq/L | 100 (2) | 98 (3)

11. Secondary Outcome: Serum CO2
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
mEq/L | 25 (1) | 25 (2)

12. Secondary Outcome: Serum Pre-albumin
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
mg/dL | 26 (7) | 26 (8)

13. Secondary Outcome: Dialysis Absences
Description: Absences out of 25 sessions
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: absences
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
absences | 0.9 (1.1) | 1.8 (2.6)

14. Secondary Outcome: Interdialytic Weight Gain
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
kg | 1.8 (1.1) | 2.4 (2.1)

15. Secondary Outcome: Vitality Score
Description: Vitality measured by SF-36 (Short Form 36 Health Survey) Questionnaire. Minimum-Maximum values 0-100, with higher scores meaning better outcomes.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 42.94 (18.30) | 42.04 (11.99)

16. Secondary Outcome: Sleep Problems Index
Description: Sleep Problems Index-II from the Medical Outcomes Study (MOS) Sleep Scale. Minimum-Maximum values 0-100, with higher scores meaning better outcomes.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 49.04 (10.2) | 43.37 (13.00)

17. Secondary Outcome: Hunger Rating
Description: Hunger rating on a visual analog scale of 0-10 cm. Higher values mean a better outcome.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meals | Control
Number analyzed (Participants) | 9 | 9
units on a scale | 1.01 (1.01) | 3.20 (1.89)

ADVERSE EVENTS:
Arm/Group | Meals | Control
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No